CLINICAL TRIAL: NCT05917886
Title: Auditory Beat Stimulation and Behavioural Variant of Frontotemporal Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Dr. Juergen Fell, Priniciple Investigator, University Hospital, Bonn
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 308/20
Record Dates: First submitted 2023-06-01; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Anxiety; bvFTD
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Patients participated in both the control and active auditory beat conditions, each lasting 1 week. Conditions were randomised across participants.
Who Masked: Participant, Care Provider
Masking Description: Participants were unaware which auditory beat stimulation condition they received in which order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monaural beat stimulation (Active Comparator): 20 min sound recording of 8Hz monaural beat
  Interventions: Other: Auditory beat stimulation: 8Hz monaural beat stimulation
- Control (Sham Comparator): 20 min sound recording of 220Hz pure sine wave
  Interventions: Other: Auditory beat stimulation: 8Hz monaural beat stimulation

INTERVENTIONS:
Other: Auditory beat stimulation: 8Hz monaural beat stimulation — Auditory beat stimulation is a reversible, non-invasive application of sound to the ears.

SUMMARY:
The goal of this study is to examine the effects of auditory beat stimulation on anxiety in patients diagnosed with bvFTD. Main aims are:

* to ascertain whether anxiety in bvFTD patients can be modulated using auditory beat stimulation
* to investigate patterns of anxiety and mind wandering in bvFTD patient population

Patients were asked to complete a number of questionnaires relating to well-being and mind wandering, as well as to listen daily to audio files of beat stimulation.

DETAILED DESCRIPTION:
Eligible patients and their caregivers were asked to give informed written consent, if they wished to participate after an initial interview. Once enrolled, they began the study by joining a consultation with their consultant neurologist and the study coordinator. Patients each received a handbook to guide them day by day during the course of the study and an mp3 player containing the auditory beat stimulation files. The handbook also contained copies of the questionnaires the patients were asked to complete at different points during the two week study (mind wandering questionnaire, State-Trait Anxiety Inventory, Beck Depression Inventory, Rogers' Happy/ Sad Face Scale). Over the course of two weeks patients completed the questionnaires and listened daily to an auditory beat stimulation or a control recording for 20 mins at home.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are the international criteria of a behavioral variant of FTD according to Raskovsky and colleagues (2011), which include:

A. Early disinhibition B. Early apathy or passivity C. Early loss of compassion or empathy D. speech or motor stereotypies E. Hyperorality and altered eating habits F. Neuropsychological profile with executive function deficits with relatively unchanged memory and visuospatial performance G. Disruption of daily living skills H. Matching imaging (cMRI, cCT, PET).

Exclusion Criteria:

* Exclusion criteria include the presence of a non-neurodegenerative psychiatric disease that can better explain the behavioral abnormalities or evidence of biomarkers with clear evidence of Alzheimer's disease or other neurodegenerative process

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Examine anxiety modulation effects of monaural beat stimulation using the State-Trait Anxiety Inventory (STAI-S and T) | 3 years
  The STAI Inventory was used to assess the patients' state (STAI-S) and trait (STAI-T) anxiety. The two subscores differentiate between transient feelings of anxiety (state anxiety), i.e. those related to a particular context like an event, and anxiety levels that are more of a personal characteristic of an individual (trait anxiety: Spielberger et al., 1983). Patients responded to 20 statements contained in each subscore, using a 4-point Likert scale (not at all: 1; a little: 2; quite: 3; very: 4). The STAI Inventory was completed at the beginning and end of each week.
Examine depression modulation effects of monaural beat stimulation using the Beck Depression Inventory | 3 years
  metric used to assess levels of depression; The BDI is a 21-item multiple-choice questionnaire (Beck et al., 1996). The BDI was used to assess symptoms of depression, and was administered at the beginning and end of each week, prior to the six-day daily course of auditory beat stimulation. The BDI is categorised into the following scoring ranges: 0-13 minimal; 14-19 mild; 20-28 moderate and 29-63 severe.
Examine mind wandering modulation effects of monaural beat stimulation using the Mind Wandering Questionnaire | 3 years
  The Mind Wandering Questionnaire is a short-form scale intended to measure the propensity to mind wander (Mrazek et al., 2013). The questionnaire consists of five items that evaluate trait levels of mind wandering. Trait mind wandering is scored across a 6-point Likert scale (1: almost never; 2: very infrequently; 3: somewhat infrequently; 4: somewhat frequently; 5: very frequently; 6: almost always). Patients completed this questionnaire, also at the beginning and end of each week.
Examine daily momentary subjective levels of anxiety, mood and pain modulation effects of monaural beat stimulation using the Mind Wandering Questionnaire | 3 years
  The Rogers' Happy/ Sad Face Scale is a visual-numeric scale that was intended to capture the momentary subjective levels of anxiety, mood and pain. Patients had to grade their feelings according to a corresponding face icon which represented a 'happy face' at the most positive end (value of 0) of the graded scale, all the way to a 'crying face' icon at the most negative end of the scale (value of 4). Patients completed this scale twice daily, once immediately prior to the auditory stimulation, and then immediately after the stimulation had concluded.

CONTACTS AND LOCATIONS:
Locations (1):
- Juergen Fell, Bonn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
All data that cannot be identified will be made available upon request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Available immediately and for the next 4 years
Access Criteria: Email and confirmation of usage.